CLINICAL TRIAL: NCT02269046
Title: A Multi-center, Randomized, Stratified, Active-controlled Trial to Evaluate the Effects of Acupuncture and Moxibustion for Hyperlipidemias
Brief Title: Acupuncture and Moxibustion for Hyperlipemia
Acronym: AMH-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Collaborators: University of British Columbia (Other); State Administration of Traditional Chinese Medicine of the People's Republic of China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LML
Record Dates: First submitted 2014-09-26; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-08

CONDITIONS: Hyperlipidemias
Keywords: acupuncture; moxibustion; hyperlipidemias; effectiveness
MeSH Terms: conditions — Hyperlipidemias | interventions — Acupuncture Therapy; Moxibustion; Simvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acupuncture and moxibustion (Experimental): * therapeutic lifestyle change
  * Group I:Juque (RN14), Tianshu (ST25, bilateral), Fenglong (ST40, bilateral), Zusanli (ST 36, bilateral), Sanyinjiao (SP6, bilateral)
  * Group II: Pishu (BL20, bilateral), Xinshu (BL15, bilateral), Ganshu (BL18, bilateral), Shenshu (BL23, bilateral)
  * Group I and II will change alternatively every other week .
  * Once per day five days per week.
  Interventions: Other: acupuncture and moxibustion; Other: Therapeutic Lifestyle Change
- Simvastatin (Active Comparator): * therapeutic lifestyle change
  * simvastatin
  * oral administration with 10mg per day
  * seven days per week for 12 weeks.
  Interventions: Drug: Simvastatin; Other: Therapeutic Lifestyle Change
- waiting list (Other): - therapeutic lifestyle change
  Interventions: Other: Therapeutic Lifestyle Change

INTERVENTIONS:
Other: acupuncture and moxibustion — Warm needling acupuncture on Fenglong (ST40, bilateral), Zusanli (ST36, bilateral), Sanyinjiao (SP6, bilateral) and Cake-seperated moxibustion on Juque (RN14), Tianshu (ST25, bilateral), Pishu (BL20, bilateral), Xinshu (BL15, bilateral), Ganshu (BL18, bilateral), Shenshu (BL23, bilateral)
  Arms: Acupuncture and moxibustion
Drug: Simvastatin — 10mg/d,p.o,12 weeks.
  Arms: Simvastatin
Other: Therapeutic Lifestyle Change — * Reduced intakes of saturated fats (<7% of total calories) and cholesterol (<200 mg per day)
  * Therapeutic options for enhancing LDL lowering
  * Weight reduction
  * Increased physical activity

SUMMARY:
The purpose of this study is to evaluate the effect of 12 weeks of acupuncture and moxibustion compared with active control, on absolute and percent change from baseline in low-density lipoprotein cholesterol (LDL-C) among those with hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Subject signed the informed consent
* Male or female ≥18 to ≤75 years of age
* Fasting TG ≤400 mg/dL
* Fasting LDL-C as determined by central laboratory on admission and meeting the following LDL-C values based on risk factor status:

  * 0-1 Risk Factor Group: LDL-C ≥160 mg/dL
  * 2+ Risk Factor Group: LDL-C ≥130 mg/dL
  * CHD or CHD risk equivalents: LDL-C ≥100 mg/dL
  * Major Risk factors: （1）Cigarette smoking;（2）Hypertension (BP ≥140/90 mmHg or on anti-hypertensive medication);（3）Low HDL cholesterol (HDL-C <40 mg/dL);（4）Family history of premature CHD (CHD in male first degree relative <55 years; CHD in female first degree relative <65 years);（5）Age (men ≥45 years; women ≥55 years)
  * CHD and CHD equivalents:（1）Other clinical forms of atherosclerotic disease (peripheral arterial disease, abdominal aortic aneurysm, and symptomatic carotid artery disease);（2）Diabetes;（3）Multiple risk factors that confer a 10-year risk for CHD >20%

Exclusion Criteria:

* CHD or CHD risk equivalent and not receiving statin therapy, with LDL-C at screening ≤99 mg/dL
* NYHA II, III or IV heart failure, or last known left ventricular ejection fraction <30%
* Uncontrolled cardiac arrhythmia, atrial fibrillation with rapid ventricular response, or not controlled supraventricular tachycardia in the past 3 months prior to randomization
* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 3 months prior to randomization
* Planned cardiac surgery or revascularization
* Type 1 diabetes or newly diagnosed type 2 diabetes or poorly controlled type 2 diabetes
* Uncontrolled hypertension defined as sitting systolic blood pressure (SBP) >160 mmHg or diastolic BP (DBP) >100 mmHg
* Subjects taken red yeast rice, niacin >200 mg/d, or omega-3 fatty acids >1000 mg/d or prescription lipid-regulating drugs other than statins or ezetimibe, such as fibrates and derivatives, or bile-acid sequestering resins in the last 6 weeks prior to LDL-C screening
* Subjects taken systemic cyclosporine, systemic steroids, vitamin A derivatives and retinol derivatives for the treatment of dermatologic conditions in the last 3 months prior to LDL-C screening
* Hyperthyroidism or hypothyroidism
* Moderate to severe renal dysfunction
* Active liver disease or hepatic dysfunction
* CK >3 times the ULN at screening or at end of lipid stabilization period, confirmed by a repeat measurement at least 1 week apart
* Known active infection or major hematologic, renal, metabolic, gastrointestinal or endocrine dysfunction in the judgment of the investigator
* Deep vein thrombosis or pulmonary embolism within 3 months prior to randomization
* Current therapeutic anticoagulation with vitamin K antagonist, heparin, low-molecular weight heparin, direct thrombin inhibitor
* Currently enrolled in another investigational device or drug study
* Female subject during pregnant or breast feeding period
* History of malignancy (except non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma)
* Known sensitivity to any of the products to be administered during dosing
* Subjects couldn't provide the written informed consent and/or comply with all required study procedures

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
low-density lipoprotein cholesterol (LDL-C) | 12 weeks
  To evaluate the effect of 12 weeks of acupuncture compared with active control, on percent change from baseline in low-density lipoprotein cholesterol (LDL-C) among those with hyperlipidemia.

SECONDARY OUTCOMES:
high-density lipoprotein cholesterol (HDL-C) | 12 weeks
total cholesterol (TC) | 12 weeks
triglyceride(TG) | 12 weeks
the rate of subjects achieving LDL-C goal | 12 weeks

OTHER OUTCOMES:
Safety | 12 weeks
  Safety summaries will include the subject incidence of adverse events, summaries of laboratory parameters (including shift tables), vital signs, and ECGs.
Adherence of acupuncture | 12 weeks
  Adherence to the treatment (adherence rate)will be calculated using formula:
  Adherence Rate = Number of Treatment Conducted/ Number of Treatment Planned

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Chang, Prof., Study Chair — Hunan University of Chinese Medicine
Locations (3):
- China (3):
  - Changsha Hospital of Chinese Medicine, Changsha, Hunan
  - Second Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan

REFERENCES:
- [Background] Yue ZH, He XQ, Chang XR, Yuan JL, Yu BS, Liu M, Fu L, Zhang L, Shang LC. The effect of herb-partition moxibustion on Toll-like receptor 4 in rabbit aorta during atherosclerosis. J Acupunct Meridian Stud. 2012 Apr;5(2):72-9. doi: 10.1016/j.jams.2012.01.005. Epub 2012 Feb 10. PMID 22483185
- [Background] Yue ZH, Yan J, Chang XR, Lin YP, Yi SX, Cao XP, Shen J. [Effects of cake-separated moxibustion on ultrastructures of endothelial cells of aorta in the rabbit of hyperlipemia]. Zhongguo Zhen Jiu. 2005 Jan;25(1):64-7. Chinese. PMID 16309161
- [Background] Xiaorong C, Jie Y, Zenghui Y, Jing S, Yaping L, Shouxiang Y, Xiangping C. Effects of medicinal cake-separated moxibustion on plasma 6-keto-PGF1alpha and TXB2 contents in the rabbit of hyperlipemia. J Tradit Chin Med. 2005 Jun;25(2):145-7. PMID 16136949
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Background] Yan X, Chen H, Gao W, Li J, Yang X, Ye P, Zhang S, Zhao D, Zhu J, Huo Y. [Consensus standpoints from expert panel of Chinese Society of Cardiology on AHA/ACC 2013 guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults]. Zhonghua Xin Xue Guan Bing Za Zhi. 2014 Apr;42(4):275-6. No abstract available. Chinese. PMID 24924450
- [Derived] Liu M, Zhang Q, Jiang S, Liu M, Zhang G, Yue Z, Chen Q, Zhou J, Zou Y, Li D, Ma M, Dai G, Zhong H, Wang Z, Chang X. Warm-needling acupuncture and medicinal cake-separated moxibustion for hyperlipidemia: study protocol for a randomized controlled trial. Trials. 2017 Jul 10;18(1):310. doi: 10.1186/s13063-017-2029-x. PMID 28693531